CLINICAL TRIAL: NCT07208045
Title: Es tu Juego: Decide Bien [It's Your Game: Keep It Real]. Cultural Adaptation, Validation, and Evaluation of the Programme for Promotion of Healthy Affective-Sexual Behaviours in Adolescents
Brief Title: Cultural Adaptation, Validation, and Evaluation of the Programme for Promotion of Healthy Affective-Sexual Behaviours in Adolescents (IYG)
Acronym: IYG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Marta Lima-Serrano, PhD, Full professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IYG2024
Record Dates: First submitted 2025-08-02; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Sexual Behavior; Sexually Transmitted Disease (STD); Condom Use; Adolescent Health; Cultural Adaptation
Keywords: sexually behaviour; sex education; adolescents; health education; cultural adaptation; evidence-based prevention; school health
MeSH Terms: conditions — Sexual Behavior; Sexually Transmitted Diseases; Health Education

STUDY DESIGN:
Intervention Model Description: The pilot effectiveness study will be conducted through a randomised community trial with a Control Group (CG) and an Intervention Group (IG). For sample size calculation, assuming an alpha risk of 0.05 and a beta risk of 0.2 in a two-sided test, 300 participants are required in the first group and 300 in the second to detect a statistically significant difference between two proportions, expected to be 0.2 for group 1 and 0.1 for group 2. A 30% loss to follow-up rate has been estimated. So it is expected to recruit 600 students in each Region, Andalusia and Catalonia. The assignment of the Control Group (CG) and Intervention Group (IG) will be carried out through simple randomisation. For allocation, each educational centre will be assigned a number, and a random number generator will be used to determine its inclusion in either the CG or IG. Participants in the CG will remain on a waiting list to receive the intervention, which will be implemented once the project is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group IYG (Experimental): The intervention group will receive the culturally adapted version of It's Your Game (IYG) educational program, which is designed to promote healthy sexual behaviors and prevent risks among adolescents.
  Interventions: Behavioral: Es tu juego: decide bien (IYG)
- Waiting list control group (No Intervention): The control group will participate in the standard sexuality and emotional education training, corresponding to the regular curriculum implemented in the educational setting. The participants in the control group will remain on a waiting list to receive the intervention, which will be implemented once the project has been completed.

INTERVENTIONS:
Behavioral: Es tu juego: decide bien (IYG) — Affective-sexual education for adolescents through an gamified online and school-based program.
  Arms: Intervention group IYG

SUMMARY:
The investigators are writing to inform participants about a study being carried out by a research group from the University of Granada and the University of Seville, in which the participant's son/daughter is invited to participate. The study has been approved by the Provincial Research Ethics Committee of Granada under code 202499906944441.

The sole intention of the investigators is to ensure that participants receive correct and sufficient information to assess and decide whether or not to give consent for the child's participation in this study. The information sheet should be read carefully, and any questions may be addressed to the investigators.

The objective of the study is to culturally adapt the program It's Your Game: Keep it Real (IYG), which aims to prevent risky sexual and affective behaviors in adolescents. The IYG program consists of 12 lessons, each lasting 45 minutes. These lessons aim to help the child identify personal norms and boundaries regarding sexuality, recognize situations that might challenge these boundaries, and develop refusal skills to maintain them. The program also covers topics such as the characteristics of healthy and unhealthy relationships, friendships, anatomy and reproduction, the social, emotional, and physical consequences of sexual activity, the consequences of teenage pregnancy and STIs, condom and contraceptive use, and communication skills.

This adaptation will involve the child completing all 12 lessons (two lessons per week over a period of six weeks) that make up the IYG program, as well as filling out a series of questionnaires. These questionnaires will allow the investigators to assess the usability of the program in Spain (including ease of use, comprehension, acceptability, as well as aspects most liked and suggestions for improvement).

Participation is entirely VOLUNTARY AND ANONYMOUS, and consent may be withdrawn at any time, without providing any explanation and without this affecting the care the child will receive in any way.

In all cases, the CONFIDENTIALITY of the data collected will be maintained in accordance with the European Union General Data Protection Regulation (GDPR) 2016/679 and the Spanish Organic Law on the Protection of Personal Data and Guarantee of Digital Rights (LOPD-GDD) 3/2018, of December 5.

Regarding the study results, these may be shared with the scientific community through presentations, conferences, and/or publications.

The investigators express appreciation in advance for cooperation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged between 11 and 14 years enrolled in compulsory secondary education (E.S.O).
* Access to a computer and internet at their educational centre.

Exclusion Criteria:

* Presence of linguistic, cognitive, or sensory barriers that prevent completion of the questionnaire
* Participation in another programme aimed at preventing affective-sexual risk behaviours.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants maintaining abstinence from oral, vaginal, and anal sex, assessed using a self-administered questionnaire adapted from It's Your Game: Keep It Real. | Baseline (Month 0), at the end of the first and second school year of implementation and the end of the following school year and end of follow-up (Month 24)
  The primary outcome will be assessed only in participants who have not initiated sexual activity at baseline. Three self-report items will be used to determine whether, since the initial assessment, the participant has initiated: Oral sex, Vaginal sex, Anal sex.
  Each question will have a dichotomous categorical response (Yes / No). The outcome will be calculated as the number and percentage of participants who respond "No" for each type of sexual activity at the end of follow-up. Data will be presented separately by study group (intervention and control) and by type of sexual activity.
  Measurement Details:
  Instrument: Structured self-administered questionnaire, culturally adapted and validated in Spanish adolescent populations during the pilot phase.
  Response format: Yes / No. Interpretation: A higher proportion of "No" responses indicates a better outcome (greater delay in the initiation of sexual activity).
  Data aggregation method: Calculation of percentages and absolute and r

CONTACTS AND LOCATIONS:
Overall Officials: Alba Sierra Yagüe, Phd Student, Principal Investigator — Catalan Institute of Health; Marta Lima Serrano, Full professor, Study Director — University of Seville; José Antonio Zafra Agea, PhD, Principal Investigator — Catalan Institute of Health; Ana Aguilar Quesada, PhD Student, Principal Investigator — San Cecilio University Hospital, Granada; María González Cano Caballero, PhD, Principal Investigator — department of Nursing, Faculty of Health Sciences, University of Granada.
Locations (1):
- IES Numancia, Barcelona, Santa Coloma de Gramenet, Spain

IPD SHARING:
Plan to Share IPD: Yes
The project will generate qualitative data (focus groups with adolescents, parents, associations, public agencies, NGOs for the cultural adaptation of the IYG program) and quantitative data (usability and pilot tests with adolescents in Andalusia and Catalonia). Data, in text and table formats, will be stored in the DIGIBUG repository (Qualified Dublin Core metadata, unique identifier, version control). They will be accessible after processing, except those protected by personal data regulations, which will be embargoed. No raw or sociodemographic data will be published. Materials will have a Creative Commons license and may be reused after project completion, with up to 3 years embargo for doctoral theses. DIGIBUG will perform backups and ensure security. Data will be pseudonymized or anonymized (AMNESIA tool) and owned by the PI, who will ensure legal and ethical compliance.
Supporting Information: SAP
Time Frame: Materials will have a Creative Commons license and may be reused after project completion, with up to 3 years embargo for doctoral theses.
Access Criteria: Raw data will only be available to the research team. Ownership of the data will rest with the project's Principal Investigator, who will ensure that no variables are transferred.

REFERENCES:
- [Background] Wiltsey Stirman S, Baumann AA, Miller CJ. The FRAME: an expanded framework for reporting adaptations and modifications to evidence-based interventions. Implement Sci. 2019 Jun 6;14(1):58. doi: 10.1186/s13012-019-0898-y. PMID 31171014
- [Background] Lucassen MF, Samra R, Brown KE, Rimes KA, Nunez-Garcia A, Wallace LM. A web-based intervention to support the mental well-being of sexual and gender minoritised adolescents: Formative evaluation of Oneself. Digit Health. 2025 Mar 13;11:20552076251321057. doi: 10.1177/20552076251321057. eCollection 2025 Jan-Dec. PMID 40093712
- [Background] Escobar-Chaves SL, Shegog R, Moscoso-Alvarez MR, Markham C, Tortolero-Luna G, Peskin M, Tortolero S. Cultural tailoring and feasibility assessment of a sexual health middle school curriculum: a pilot test in Puerto Rico. J Sch Health. 2011 Aug;81(8):477-84. doi: 10.1111/j.1746-1561.2011.00617.x. PMID 21740433
- [Background] Virzi RA. Refining the Test Phase of Usability Evaluation: How Many Subjects Is Enough? Human Factors: The Journal of the Human Factors and Ergonomics Society. 1992; 1; 34(4): 457-68. https://2024.sci-hub.box/3857/2afb54700f6961ae637e388c3f96891c/virzi1992.pdf
- [Background] Vargas-Martinez AM, Guillen-Martinez D, Domingo Perez T, Soilan Enriquez A, Zafra-Agea JA, Hoyos Cillero I, Lima-Serrano M, Tarrino-Concejero L. Analysis of the management function of the school nurse in Spain: use of records and interaction with primary care, the educational community and other institutions. Enferm Clin (Engl Ed). 2025 Sep-Oct;35(5):502200. doi: 10.1016/j.enfcle.2025.502200. Epub 2025 May 22. PMID 40412717
- [Background] Agyei FB, Kaura DK, Bell JD. Parent-adolescent sexual and reproductive health information communication in Ghana. Reprod Health. 2025 Feb 19;22(1):25. doi: 10.1186/s12978-025-01961-y. PMID 39972503
- [Background] Mukanga B, Dlamini SB, Taylor M. Cultural appropriateness of a comprehensive sexuality education programme. Implications for programme adaptation and implementation in Zambia. Sex Educ. 2025; 3;25(5): 631-46. https://doi.org/10.1080/14681811.2024.2367761
- [Background] Kitzinger J. Qualitative research. Introducing focus groups. BMJ. 1995 Jul 29;311(7000):299-302. doi: 10.1136/bmj.311.7000.299. PMID 7633241
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] Lee SD, Iott B, Banaszak-Holl J, Shih SF, Raj M, Johnson KE, Kiessling K, Moore-Petinak N. Application of Mixed Methods in Health Services Management Research: A Systematic Review. Med Care Res Rev. 2022 Jun;79(3):331-344. doi: 10.1177/10775587211030393. Epub 2021 Jul 12. PMID 34253078
- [Background] Leech N, Onwuegbuzie A. Guidelines for conducting and reporting mixed research in the field of counseling and beyond. Journal of Counseling and Development. 2010; 88(1): 61-9. doi: 10.1002/j.1556-6678.2010.tb00151.x
- [Background] Muheriwa-Matemba S, Crooks N, Hall H et al. 156. Fostering Young Adolescent Engagement in Sexual Health Research: A Youth-Led Community-Based Participatory Research in Western NY. Journal of Adolescent Health. 2025; 76(3): S81. doi: 10.1016/j.jadohealth.2024.11.172
- [Background] Meherali S, Munro S, Puinean G, Salami B, Wong JP, Vandermorris A, Benoit JRA, Flicker S, Okeke-Ihejirika P, Stroulia E, Norman WV, Scott SD. Co-designing a Sexual Health App With Immigrant Adolescents: Protocol for a Qualitative Community-Based Participatory Action Research Study. JMIR Res Protoc. 2023 Mar 22;12:e45389. doi: 10.2196/45389. PMID 36947124
- [Background] Kachingwe ON, Lewis Q, Offiong A, Smith BD, LoVette A, Powell TW. Using the intervention mapping for adaption framework to adapt an evidence-based sexual health intervention for youth affected by trauma. BMC Public Health. 2023 Jun 1;23(1):1052. doi: 10.1186/s12889-023-15984-2. PMID 37264451
- [Background] Resnicow K, Baranowski T, Ahluwalia JS, Braithwaite RL. Cultural sensitivity in public health: defined and demystified. Ethn Dis. 1999 Winter;9(1):10-21. PMID 10355471
- [Background] Bernal G, Bonilla J, Bellido C. Ecological validity and cultural sensitivity for outcome research: issues for the cultural adaptation and development of psychosocial treatments with Hispanics. J Abnorm Child Psychol. 1995 Feb;23(1):67-82. doi: 10.1007/BF01447045. PMID 7759675
- [Background] Corpus-Espinosa C, Mac Fadden I, Del Carmen Torrejon-Guirado M, Lima-Serrano M. Exploring Cultural Adaptations: A Scoping Review on Adolescent Mental Health and Substance Use Prevention Programs. Prev Sci. 2025 Feb;26(2):204-221. doi: 10.1007/s11121-025-01779-x. Epub 2025 Jan 31. PMID 39888521
- [Background] Flay BR, Petraitis J. The Theory of Triadic Influence: A New Theory of Health Behavior With Implications for Preventive Interventions. Advances in Medical Sociology 1994. https://www.researchgate.net/publication/224942196_The_Theory_of_Triadic_Influence_A_New_Theory_of_Health_Behavior_With_Implications_for_Preventive_Interventions
- [Background] Perry CL. Creating health behavior change: How to develop community-wide programs for youth. Sage Publications, editor. Thousand Oaks, California, USA; 1999.
- [Background] Komro KA, Perry CL, Williams CL, Stigler MH, Farbakhsh K, Veblen-Mortenson S. How did Project Northland reduce alcohol use among young adolescents? Analysis of mediating variables. Health Educ Res. 2001 Feb;16(1):59-70. doi: 10.1093/her/16.1.59. PMID 11252284
- [Background] Bandura A. Social foundations of thought and action: a social cognitive theory. Englewood Cliffs: Prentice Hall; 1986.
- [Background] Lima-Serrano M, Barrera-Villalba C, Mac-Fadden I, Mesters I, de Vries H. Alerta Cannabis: A Tailored-Computer Web-Based Program for the Prevention of Cannabis Use in Adolescents: A Cluster-Randomized Controlled Trial Protocol. BMC Nurs. 2024 Apr 10;23(1):239. doi: 10.1186/s12912-024-01889-x. PMID 38600496
- [Background] Shegog R, Craig Rushing S, Gorman G, Jessen C, Torres J, Lane TL, Gaston A, Revels TK, Williamson J, Peskin MF, D'Cruz J, Tortolero S, Markham CM. NATIVE-It's Your Game: Adapting a Technology-Based Sexual Health Curriculum for American Indian and Alaska Native youth. J Prim Prev. 2017 Apr;38(1-2):27-48. doi: 10.1007/s10935-016-0440-9. PMID 27520459
- [Background] Shegog R, Peskin MF, Markham C, Thiel M, Karny E, Addy RC, Johnson KA, Tortolero S. It's Your Game-Tech: Toward Sexual Health in the Digital Age. Creat Educ. 2014 Aug;5(15):1428-1447. doi: 10.4236/ce.2014.515161. PMID 25705561
- [Background] Peskin MF, Shegog R, Markham CM, Thiel M, Baumler ER, Addy RC, Gabay EK, Emery ST. Efficacy of It's Your Game-Tech: A Computer-Based Sexual Health Education Program for Middle School Youth. J Adolesc Health. 2015 May;56(5):515-21. doi: 10.1016/j.jadohealth.2015.01.001. Epub 2015 Mar 1. PMID 25739520
- [Background] Markham CM, Tortolero SR, Peskin MF, Shegog R, Thiel M, Baumler ER, Addy RC, Escobar-Chaves SL, Reininger B, Robin L. Sexual risk avoidance and sexual risk reduction interventions for middle school youth: a randomized controlled trial. J Adolesc Health. 2012 Mar;50(3):279-88. doi: 10.1016/j.jadohealth.2011.07.010. Epub 2011 Oct 7. PMID 22325134
- [Background] Tortolero SR, Markham CM, Peskin MF, Shegog R, Addy RC, Escobar-Chaves SL, Baumler ER. It's Your Game: Keep It Real: delaying sexual behavior with an effective middle school program. J Adolesc Health. 2010 Feb;46(2):169-79. doi: 10.1016/j.jadohealth.2009.06.008. Epub 2009 Aug 18. PMID 20113923

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-29): https://cdn.clinicaltrials.gov/large-docs/45/NCT07208045/Prot_SAP_000.pdf
  • Informed Consent Form: Infomed consent (2025-05-29): https://cdn.clinicaltrials.gov/large-docs/45/NCT07208045/ICF_001.pdf